CLINICAL TRIAL: NCT00074633
Title: Evaluating "Health at Every Size"(HAES) as an Alternative Obesity Treatment Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: University of California, Davis (Other); United States Department of Agriculture (USDA) (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBFRETTO (completed)
Record Dates: First submitted 2003-12-17; First posted 2003-12-19 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Hypercholesterolemia; Hypertension; Depression; Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes; Self-Esteem
MeSH Terms: conditions — Hypercholesterolemia; Hypertension; Depression; Diabetes Mellitus, Type 2 | interventions — Diet

INTERVENTIONS:
Behavioral: Health at Every Size (HAES)
Behavioral: Diet (Traditional, moderate energy restriction)

SUMMARY:
Increasingly more individuals are trying to lose weight. Indeed, many women, regardless of their size, experience a life-long battle and preoccupation with their weight. Despite the attention to weight and the increase in diet behavior, the incidence of obesity continues to rise. There is little data to show improved long term success for the majority of participants who engage in weight loss behaviors.

The specific aim is to improve the psychological and metabolic health of obese women with a history of chronic dieting through encouraging "Health at Every Size" (HAES). This treatment model emphasizes "intutitive eating," i.e., internal regulation of eating (responding to cues of hunger, appetite and satiety). The HAES model is being compared to the current standard of care in obesity treatment, energy restriction dieting, which encourages cognitive control of eating and weight reduction.

ELIGIBILITY:
* Caucasian;
* female;
* age 30-45 years;
* Body Mass Index (BMI)>30 m/kg2;
* non-smoker;
* not pregnant or lactating;
* Restraint Scale (Herman and Polivy, 1988) score >15, indicating a history of chronic dieting;
* no recent myocardial infarction;
* no active neoplasms, Type 1 diabetes or insulin-dependent Type 2 diabetes, nor history of cerebrovascular or renal disease.

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79
Dates: Start 2000-01

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Nutrition Department, University of California, Davis, Davis, California
  - Western Human Nutrition Research Center, Davis, California

REFERENCES:
- [Background] Bacon L, Keim NL, Van Loan MD, Derricote M, Gale B, Kazaks A, Stern JS. Evaluating a 'non-diet' wellness intervention for improvement of metabolic fitness, psychological well-being and eating and activity behaviors. Int J Obes Relat Metab Disord. 2002 Jun;26(6):854-65. doi: 10.1038/sj.ijo.0802012. PMID 12037657